CLINICAL TRIAL: NCT00341198
Title: Confirmation of Systemic Autoimmune Diseases in the Agricultural Health Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902166; 02-E-N166
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-12

CONDITIONS: Autoimmune Disease
Keywords: Rheumatoid Arthritis; Lupus; Scleroderma; Sjogren's Syndrome; Farming; Autoimmune Disease; Exposure
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Rheumatoid; Scleroderma, Diffuse; Sjogren's Syndrome

SUMMARY:
Autoimmune diseases may involve nearly any organ and are characterized by abnormal activation or response of certain cells. Evidence suggests that farm work, exposure to silica from farming activities and exposure to pesticides may contribute to the development of autoimmune disease. Associations between autoimmune diseases and farming, however, have not been extensively investigated, and exposure data in the currently available studies are extremely limited.

One of the major challenges in conducting population-based research on autoimmune diseases is case ascertainment. Self-report of previous diagnosis has proven to be unreliable. This protocol outlines a strategy to confirm self-reported diagnoses of systemic autoimmune diseases (rheumatoid arthritis, systemic lupus erythematosus, scleroderma, and Sjogren syndrome) within the Agricultural Health Study group (AHS; a group of licensed pesticide applicators and spouses who completed a questionnaire). The confirmed cases will constitute a refined case group to allow analyses of pesticides and other farming-related exposures as possible risk factors for these diseases using data that have already been collected.

Subjects will be selected from participants in the AHS who reported one of the diseases being studied. A short telephone interview will be conducted with participants, who will be requested to provide written consent for review of information from medical records. To confirm the self-diagnosis, participants' physicians will be contacted. Specific information will be requested in the form of a checklist. Responses will be reviewed for evidence of diagnosis and classified as confirmed, probable, physician-diagnosed, or unconfirmed.

Secondary objectives of this study are to:

* assess the correct interpretation of conflicting self-reports that are provided at two different times.
* evaluate the usefulness of specific questions that could potentially be used in future studies to validate self-reported cases of rheumatoid arthritis in men.

DETAILED DESCRIPTION:
Farming-related exposures (including pesticides and silica) may contribute to the etiology of autoimmune diseases. However, associations between autoimmune diseases and farming have not been extensively investigated, and exposure data in the currently available studies is extremely limited. One of the major challenges in conducting population-based research on autoimmune diseases is case ascertainment. Self-report of previous diagnosis has been shown to be very unreliable. This protocol outlines a strategy to confirm self-reported diagnoses of systemic autoimmune diseases (rheumatoid arthritis, systemic lupus erythematosus, scleroderma, and Sjogren syndrome) within the Agricultural Health Study (AHS) cohort. The confirmed cases will constitute a refined case group to allow etiologic analyses of pesticides and other farming-related exposures as possible risk factors for these diseases using data that have already been collected. The codes can also be used in a nested case-control study that could be designed to collect additional exposure data (for example, on silica-related exposures).

ELIGIBILITY:
* INCLUSION CRITERIA:

Agricultural workers and their spouses.

EXCLUSION CRITERIA:

Children will not be included.

There are no exclusions based on ethnicity or race.

Participants who are unable to complete a telephone interview because of chronic illness (including cognitive impairment) or language or hearing difficulties will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2002-04-02; Study Completion 2006-12-12

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Battelle Centers for Public Health Research and Evaluation, Durham, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Jubault V, Penfornis A, Schillo F, Hoen B, Izembart M, Timsit J, Kazatchkine MD, Gilquin J, Viard JP. Sequential occurrence of thyroid autoantibodies and Graves' disease after immune restoration in severely immunocompromised human immunodeficiency virus-1-infected patients. J Clin Endocrinol Metab. 2000 Nov;85(11):4254-7. doi: 10.1210/jcem.85.11.6988. PMID 11095463